CLINICAL TRIAL: NCT06383871
Title: An Open, Multicenter Phase I Study of Safety, Tolerability, Pharmacokinetics, and Efficacy of HRS-7058 Monotherapy in Patients With Advanced Solid Tumour With KRAS G12C Mutation
Brief Title: A Phase I Clinical Study of HRS-7058 in Patients With Advanced Malignant Tumour
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7058-101
Record Dates: First submitted 2024-04-19; First posted 2024-04-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Advanced Malignant Tumour

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-7058 (Experimental)
  Interventions: Drug: HRS-7058 capsule/ HRS-7058 tablet

INTERVENTIONS:
Drug: HRS-7058 capsule/ HRS-7058 tablet — HRS-7058 capsule/ HRS-7058 tablet

SUMMARY:
This study is a multicentre, open phase I clinical study of dose escalation, dose extension and efficacy extension of HRS-7058 in subjects with advanced malignant tumour. To evaluate the safety, tolerability, pharmacokinetics and efficacy of HRS-7058.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects gave informed consent to the study before participating in, and voluntarily signed informed consent;
2. 18 to 75 years old (including both ends), gender is not limited;
3. Subjects with locally advanced or metastatic solid tumour confirmed by histopathology;
4. Having at least one evaluable or measurable lesion according to the solid tumour response Evaluation Criteria (RECIST 1.1);
5. ECOG Performance Status of 0 or 1;
6. The expected survival time is more than 3 months;
7. Be able to ingest drugs and be able to comply with trial and follow-up procedures;
8. Adequate bone marrow and organ function;
9. Fertile women must agree to abstain from sex (abstaining from heterosexual intercourse) or use a highly effective method of contraception for at least one week from the time they sign an informed consent form until the last dose of the study drug. The blood HCG test must be negative within 7 days before the start of the study treatment, and must be non-lactating;
10. For male patients whose partner is a woman of reproductive age, they must agree to abstain from sex for at least one week from signing the informed consent until the last dose of the study drug, or to use a highly effective method of contraception.

Exclusion Criteria:

1. Accompanied by untreated or active central nervous system (CNS) tumour metastasis;
2. Had other malignancies within five years prior to first use of the investigational drug;
3. With severe cardiovascular and cerebrovascular disease；
4. Refractory nausea, vomiting, or other gastrointestinal disorders that affect the use of oral medications;
5. The presence of uncontrolled pleural, abdominal or pericardial effusion;
6. Severe infection within 4 weeks prior to initiation of study treatment;
7. History of immune deficiency;
8. The adverse reactions of previous anti-tumour therapy have not recovered to CTCAE ≤ grade 1;
9. Antitumor therapy such as chemotherapy, biotherapy, targeted therapy, immunotherapy, or other unmarketed investigational drug therapy within 4 weeks prior to initial use of the investigational drug;
10. Had undergone major organ surgery within 4 weeks prior to the first use of the study drug;
11. Women who are pregnant, breastfeeding, or who plan to become pregnant within one week of their last use of the study drug during the study period;
12. Known allergies and contraindications to the investigational drug or any of its components;
13. In the investigator's judgment, the subjects had other factors that could have affected the study results or led to the forced termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | From the beginning of first patient in (FPI) to the end of dose escalation phase up to approximately 10 months
maximum tolerated dose (MTD) | From the beginning of first patient in (FPI) to the end of dose escalation phase up to approximately 10 months
Phase II recommended dose (RP2D) | From the beginning of first patient in (FPI) to the end of dose escalation phase up to approximately 10 months
Safety endpoints: adverse events (AE) | From the beginning of first patient in (FPI) to the end of study up to approximately 21 months]

SECONDARY OUTCOMES:
Efficacy endpoints: Objective response rate (ORR) assessed based on RECIST v1.1 criterion | From the beginning of first patient in (FPI) to the end of study up to approximately 21 months
Efficacy endpoints: duration of response (DoR) assessed based on RECIST v1.1 criterion | From the beginning of first patient in (FPI) to the end of study up to approximately 21 months
Efficacy endpoints: disease control rate (DCR) assessed based on RECIST v1.1 criterion | From the beginn ing of first patient in (FPI) to the end of study up to approximately 21 months
Efficacy endpoints: progression-free survival (PFS) assessed based on RECIST v1.1 criterion | From the beginn ing of first patient in (FPI) to the end of study up to approximately 21 months
Efficacy endpoints: overall survival (OS) | From the beginn ing of first patient in (FPI) to the end of study up to approximately 21 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided